CLINICAL TRIAL: NCT05839236
Title: COVID-19 Vaccination Detoxication in Low Density Lipoprotein Cholesterol
Brief Title: COVID-19 Vaccination Detoxification in LDL-C
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yang I. Pachankis (Individual)
Responsible Party: Sponsor-Investigator, Yang I. Pachankis, Researcher, Pachankis, Yang I., M.D.
Organization: Pachankis, Yang I., M.D. (Individual)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SARSCoVVAXDetox
Record Dates: First submitted 2023-05-01; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Stress Syndrome; COVID-19 Vaccine Adverse Reaction; COVID-19-Associated Thromboembolism; COVID-19 Post-Intensive Care Syndrome; COVID-19-Associated Stroke; COVID-19 Respiratory Infection
Keywords: COVID-19; SARS-CoV-2; Low Density Lipoprotein Cholesterol; sebum; immune reflex; immunology; immune deficiency; immune regulation; detoxification
MeSH Terms: conditions — COVID-19 stress syndrome; COVID-19 post-intensive care syndrome; COVID-19; Immunologic Deficiency Syndromes | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LDL-C Detox (Experimental): The participant is continued from the trial NCT05711810. The follow-up study is separately registered for the etiological evidence from vaccine poisoning.
  With the prior study's angiotensin-converting enzyme receptor inhibition therapy reaching desired power level and outcome, the participant's blood pressure. has dropped to normal range in a steady state without signs of sudden death risks.
  The separate study defines the treatment medicines in NCT05711810 as rescue medicines for discretions, and experiments with Atorvastatin Calcium Tablets with 20 mg per day, and Chinese herb compounded Anti-Viral Granules 12 g (total) in 3 times per day.
  The main ingredients for Anti-Viral Granules are the roots of Isatis indigotica L., Forsythia suspensa, Gypsum, Common Anemarrhena, Reed Rhizome, Rehmannia glutinosa, Patchouli, Tatarinow Sweerflag Rhizome, and Curcuma aromatica. They're mixed with dextrin, Sodium cyclamate, patchouli oil, peppermint oil, and angelica dahurica tincture.
  Interventions: Combination Product: Atorvastatin Calcium Tablets

INTERVENTIONS:
Combination Product: Atorvastatin Calcium Tablets — The intervention observes the effects of the medicines on the participant's health without the continued interventions on blood pressure. Rescue medicines will be used once if the blood pressure rise again beyond the healthy range.
  Other Names: Anti-Viral Granules

SUMMARY:
The study hypothesizes that SARS-CoV-2 vaccination poisoning hibernates in human host in Low Density Lipoprotein Cholesterol (LDL-C). The clinical trial is a follow-up from the intervention trial with NCT number NCT05711810. It tests the use of Atorvastatin Calcium Tablets for detoxification and prevention of blood acidification, and the use of the Chinese herb compounded Anti-Viral Granules for the detoxification in the endocrine system.

ELIGIBILITY:
Inclusion Criteria:

* People who received COVID-19 vaccinations, or experiencing long-COVID.

Exclusion Criteria:

* People with moderate and severe liver dysfunctions.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Total Cholesterol Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication. It is hypothesized that total cholesterol levels indicate to the initial acidification for SARS-CoV-2 viral entry through vaccines with the degeneration of lipids.
Triglycerides Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication. It is hypothesized that triglycerides levels indicate to the initial acidification for SARS-CoV-2 viral entry through vaccines.
HDL-C Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
LDL-C Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication. It is hypothesized that SARS-CoV-2 hibernating viruses and viral proteins are hidden in the LDL-C.
Apolipoprotein A-I Change | 30 days
Apolipoproteina B Change | 30 days
Lipopoliproteina (a) Change | 30 days
Eosinophil Absolute Number Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Eosinophil Percentage Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Basophil Absolute Number Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Basophil Percentage Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Mean Corpuscular Volume Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Mean Corpuscular Hemoglobin Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Mean Corpuscular Hemoglobin Concentration Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Red cell Distribution Width Coefficient of Variation Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Red cell Distribution Width Standard Deviation Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Plateletcrit Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Platelet Distribution Width Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.
Mean Platelet Volume Change | 30 days
  The baseline characteristics is set at the beginning of the trial, with its rate of change metrified from initial intoxication.

SECONDARY OUTCOMES:
Heart Rate Change | 4 hours
  The blood pressure change will be compared with the baseline characteristics for observation on the risks of rebound to the previous intervention. Type I error testing defines Systolic & Diastolic Blood Pressure and heart rate as incremented. Heart rate variance indicates to immune responses.
Systolic Blood Pressure Change | 4 hours
  The blood pressure change will be compared with the baseline characteristics for observation on the risks of rebound to the previous intervention. Type I error testing defines Systolic & Diastolic Blood Pressure and heart rate as incremented. SBP variance indicates to infection activities.
Diastolic Blood Pressure Change | 4 hours
  The blood pressure change will be compared with the baseline characteristics for observation on the risks of rebound to the previous intervention. Type I error testing defines Systolic & Diastolic Blood Pressure and heart rate as incremented. DBP variance indicates to immune attack activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Residential Address, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data collected will be deidentified and shared on Zenodo with the same entry currently assigned the doi: 10.5281/zenodo.7856000.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 60 days.
Access Criteria: Study protocol with SAP and ICF will be shared at the early phase of the trial. Clinical Study Report will be shared either as a link to publication or directly on the system.

REFERENCES:
- [Background] Smith KR, Thiboutot DM. Thematic review series: skin lipids. Sebaceous gland lipids: friend or foe? J Lipid Res. 2008 Feb;49(2):271-81. doi: 10.1194/jlr.R700015-JLR200. Epub 2007 Nov 1. PMID 17975220
- [Background] Lovaszi M, Szegedi A, Zouboulis CC, Torocsik D. Sebaceous-immunobiology is orchestrated by sebum lipids. Dermatoendocrinol. 2017 Oct 17;9(1):e1375636. doi: 10.1080/19381980.2017.1375636. eCollection 2017. PMID 29484100
- [Background] Zouboulis CC, Coenye T, He L, Kabashima K, Kobayashi T, Niemann C, Nomura T, Olah A, Picardo M, Quist SR, Sasano H, Schneider MR, Torocsik D, Wong SY. Sebaceous immunobiology - skin homeostasis, pathophysiology, coordination of innate immunity and inflammatory response and disease associations. Front Immunol. 2022 Nov 10;13:1029818. doi: 10.3389/fimmu.2022.1029818. eCollection 2022. PMID 36439142
- [Background] Sorgato MC, Ferguson SJ, Kell DB, John P. The protonmotive force in bovine heart submitochondrial particles. Magnitude, sites of generation and comparison with the phosphorylation potential. Biochem J. 1978 Jul 15;174(1):237-56. doi: 10.1042/bj1740237. PMID 212021
- [Background] EVANS MC. THE PHOTO-OXIDATION OF SUCCINATE BY CHROMATOPHORES OF RHODOSPIRILLUM RUBRUM. Biochem J. 1965 Jun;95(3):661-8. doi: 10.1042/bj0950661. PMID 14342500
- [Background] Mackey K, Ayers CK, Kondo KK, Saha S, Advani SM, Young S, Spencer H, Rusek M, Anderson J, Veazie S, Smith M, Kansagara D. Racial and Ethnic Disparities in COVID-19-Related Infections, Hospitalizations, and Deaths : A Systematic Review. Ann Intern Med. 2021 Mar;174(3):362-373. doi: 10.7326/M20-6306. Epub 2020 Dec 1. PMID 33253040
- [Background] Mathur R, Rentsch CT, Morton CE, Hulme WJ, Schultze A, MacKenna B, Eggo RM, Bhaskaran K, Wong AYS, Williamson EJ, Forbes H, Wing K, McDonald HI, Bates C, Bacon S, Walker AJ, Evans D, Inglesby P, Mehrkar A, Curtis HJ, DeVito NJ, Croker R, Drysdale H, Cockburn J, Parry J, Hester F, Harper S, Douglas IJ, Tomlinson L, Evans SJW, Grieve R, Harrison D, Rowan K, Khunti K, Chaturvedi N, Smeeth L, Goldacre B; OpenSAFELY Collaborative. Ethnic differences in SARS-CoV-2 infection and COVID-19-related hospitalisation, intensive care unit admission, and death in 17 million adults in England: an observational cohort study using the OpenSAFELY platform. Lancet. 2021 May 8;397(10286):1711-1724. doi: 10.1016/S0140-6736(21)00634-6. Epub 2021 Apr 30. PMID 33939953
- [Background] Zhao M, Luo Z, He H, Shen B, Liang J, Zhang J, Ye J, Xu Y, Wang Z, Ye D, Wang M, Wan J. Decreased Low-Density Lipoprotein Cholesterol Level Indicates Poor Prognosis of Severe and Critical COVID-19 Patients: A Retrospective, Single-Center Study. Front Med (Lausanne). 2021 May 26;8:585851. doi: 10.3389/fmed.2021.585851. eCollection 2021. PMID 34124081
- [Background] Knox PP, Lukashev EP, Korvatovskii BN, Seifullina NK, Goryachev SN, Allakhverdiev ES, Paschenko VZ. Effect of Dipyridamole on Membrane Energization and Energy Transfer in Chromatophores of Rba. sphaeroides. Biochemistry (Mosc). 2022 Oct;87(10):1138-1148. doi: 10.1134/S0006297922100078. PMID 36273882
- [Background] DE Flora S, Balansky R, LA Maestra S. Antioxidants and COVID-19. J Prev Med Hyg. 2021 Jun 5;62(1 Suppl 3):E34-E45. doi: 10.15167/2421-4248/jpmh2021.62.1S3.1895. eCollection 2021 Mar. Italian. PMID 34622082
- [Background] Seneff S, Kyriakopoulos AM, Nigh G, McCullough PA. A Potential Role of the Spike Protein in Neurodegenerative Diseases: A Narrative Review. Cureus. 2023 Feb 11;15(2):e34872. doi: 10.7759/cureus.34872. eCollection 2023 Feb. PMID 36788995
- [Background] Salih RQ, Salih GA, Abdulla BA, Ahmed AD, Mohammed HR, Kakamad FH, Salih AM. False-positive HIV in a patient with SARS-CoV-2 infection; a case report. Ann Med Surg (Lond). 2021 Nov;71:103027. doi: 10.1016/j.amsu.2021.103027. Epub 2021 Nov 6. PMID 34777794
- [Background] Yang IP. Theoretical Strategies in SARS-CoV-2 Human Host Treatment. Journal of Clinical and Medical Images. 2023; 6(28).
- [Background] Yang IP. Cardiac Transfer of SARS-CoV-2 Spike Protein Circulation Techniques - Medicine Induced Hemodialysis on "Vaccinated" Immune Attacks. Biomedical Science and Clinical Research. 2023; 2(1): 86-93.
- Available data/document: Individual Participant Data Set: 10.5281/zenodo.7883407 — https://doi.org/10.5281/zenodo.7856000 — The identifier is reserved and the repository team is helping solving the technical issues in updating the data with the renewed identifier.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT05839236/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05839236/ICF_001.pdf